CLINICAL TRIAL: NCT03530904
Title: Comparison Between Early and Late Post-operative Mobilization Following Implantation of Cardiac Pacemaker or Defibrillator
Brief Title: Comparison Between Early and Late Mobilization After Cardiac Device Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Asaf Danon, Principal investigator, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-17-0015-CTIL
Record Dates: First submitted 2018-04-02; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pacemaker, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early mobilization after cardiac device implantation (Active Comparator): mobilization after 4 hours
  Interventions: Other: mobilization
- Late mobilization after cardiac device implantation (Active Comparator): Mobilization after 24 hours
  Interventions: Other: mobilization

INTERVENTIONS:
Other: mobilization — Early mobilization after CIED implantation

SUMMARY:
Mobilization after cardiac implantable electronic devices (CIED) implantation is highly variable between centers, some discharging home after 3-4 hours while others request bed restriction for 24 hours. Concern about lead dislodgements due to early mobilization are probably not justified. Bed restriction may result in considerable inconvenience to the patients.

DETAILED DESCRIPTION:
Mobilization after cardiac implantable electronic devices (CIED) implantation is highly variable between centers, some discharging home after 3-4 hours while others request bed restriction for 24 hours. Concern about lead dislodgements due to early mobilization are probably not justified. Bed restriction may result in considerable inconvinience to the patients.

Patients will be randomally assigned to early mobilization (after 4 hours) or bed restriction till the morning after the procedure.

Primary outcome: lead malfunction, patients' satisfaction

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing device implantation and are hemodynamically stable

Exclusion Criteria:

* hemodincamically unstable
* patient's request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Lead dislodgement | one month
  incidence of device lead dislodgement

SECONDARY OUTCOMES:
Patients' comfort level | one month
  comfort level based on immobilization comfort questionnaire

IPD SHARING:
Plan to Share IPD: No